CLINICAL TRIAL: NCT03626038
Title: A.L.P.S. Proximal Humerus Plating System Post-Market Clinical Follow-up Study
Brief Title: Post Market Clinical Follow-up (PMCF) Study of the A.L.P.S. Proximal Humerus Plating System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2017-59T
Record Dates: First submitted 2018-07-23; First posted 2018-08-10 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-Traumatic Arthritis; Psoriatic Arthritis; Proximal Humeral Fracture
Keywords: Trauma; Medical Device; Performance; Safety; Proximal Humeral Fracture
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic; Shoulder Fractures; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients who receive the A.L.P.S. Prox. Humerus Plating Sys. (Experimental): Subjects in need of proximal humerus fracture fixation who met the inclusion/exclusion criteria and received the A.L.P.S. Proximal Humerus Plating System.
  Subjects can be enrolled prospectively or retrospectively as indicated in the protocol.
  Interventions: Device: A.L.P.S. Proximal Humerus Plating System

INTERVENTIONS:
Device: A.L.P.S. Proximal Humerus Plating System — Anatomically contoured, locking plates that can be customized intra-operatively, multidirectional screws allow for stable fixation for a wide variety of patients.

SUMMARY:
This study is a multicenter, prospective, non-randomized, non-controlled post-market clinical follow-up study. The primary objective of this study is to confirm the safety and performance of the A.L.P.S. Proximal Humerus Plating System applied in proximal humerus fracture treatment.

DETAILED DESCRIPTION:
The A.L.P.S. Proximal Humerus Plating System was developed to provide another surgical option for proximal humerus fracture fixation. The aim of the A.L.P.S. Proximal Humerus Plating System is to provide increased fracture stability while simultaneously increasing range of motion and decreasing the likelihood of screw perforation.

A minimum of 7 and maximum of 10 sites globally will be involved in this study. This number of clinical sites will allow for a better generalization of study data as well as allow for consistency to be developed across multiple regions. 135 implants will be included into the study. Each site will be allowed to enroll 27 humeri. Enrollment is competitive. All potential study subjects will be required to participate in the Informed Consent process.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must have a primary proximal humerus fracture (Orthopaedic Trauma Association/ American Orthopedic 11-A, B, C) requiring surgical intervention and be eligible for fixation by plate and screws.
* Patients with failed conservative treatment within 3 weeks since injury.
* Patient must be able and willing to complete the protocol required follow-up.
* Patient must have a signed Institutional Review Board/Ethics Committee approved informed consent.
* Patient must be in a good nutritional state

Exclusion Criteria:

* Delay of surgery for more than 3 weeks.
* Tumor induced fractures
* Patient is a prisoner.
* Pregnancy/ breast feeding
* Patient is a current alcohol or drug abuser.
* Patient has a mental or neurologic condition that will not allow for proper informed consent and/or participation in follow-up program.
* Patient has an active infection.
* Patient conditions including limitations in blood supply, obesity, or insufficient quantity or quality of bone stock.
* Patient is sensitive to foreign body material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Re-operation | 1 year
  Re--operation within the first year post-initial surgery due to screw perforation of the humeral head, secondary displacement or impingement to relieve pain and/or improve function.

SECONDARY OUTCOMES:
Clinical efficacy of the device is assessed using the American Shoulder and Elbow Surgeon Patient Questionnaire | 2 years
  Pain, function and activities of daily living are measured. The American Shoulder and Elbow Surgeon (ASES) scale is 0 to 100. 100 is the highest score and indicates the greatest function while 0 is the lowest score.
Shoulder range of motion measurement | 2 years
  Shoulder range of motion is assessed in degrees of directional movement. This will be measured during a physical exam by the investigator. Values measured include active and passive range of motion.
Clinical performance of the device is assessed using x-ray capture | 2 years
  X-ray capture will be used to analyze fracture healing

CONTACTS AND LOCATIONS:
Locations (7):
- Foundation for Orthopaedic Research & Education, Tampa, Florida, United States
- Sydney Adventist Hospital, Wahroonga, New South Wales, Australia
- The Research Institute of McGill University Health Centre, Montreal, Quebec, Canada
- South Korea (3):
  - Korea University Anam Hospital, Seoul, Seoul
  - Hallym University Kangnam Sacred Hearth Hospital, Seoul, Seoul
  - Inje University Seoul Paik Hospital, Seoul, Seoul
- Bone and Motion Training and Research Foundation, Granges-Paccot, Granges-Paccot, Switzerland

IPD SHARING:
Plan to Share IPD: No